CLINICAL TRIAL: NCT06209840
Title: The Effect of Music Therapy on Upper Extremity Functions and Quality Of Life in Individuals With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Nezehat Özgül, Lecturer, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AYBU-NOUNLER-001
Record Dates: First submitted 2024-01-06; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy; Hemiplegic Cerebral Palsy; Music Therapy
Keywords: Cerebral Palsy; Music Therapy; Upper Extremity; Quality of Life
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups; Population Groups; Music Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Classical physiotherapy program will be applied for gross motor functions and upper extremity functions.
  Interventions: Other: Control Group
- Study (Music) Group (Experimental): In addition to the classical physiotherapy program for gross motor functions, will be applied in the Neuro-Creative Music Therapy (NCMT) program for upper extremity.
  Interventions: Other: Study (Music) Group

INTERVENTIONS:
Other: Control Group — The session is 50 minutes long and consists of 20 minutes of classical physiotherapy for gross motor functions and 30 minutes of classical physiotherapy for the upper extremity. A total of 16 sessions will be applied 2 days a week for 8 weeks.
  Other Names: Classical Physiotherapy
  Arms: Control Group
Other: Study (Music) Group — The session is 50 minutes long and consists of 20 minutes of classical physiotherapy for gross motor functions and 30 minutes of music therapy for the upper extremity. A total of 16 sessions will be applied 2 days a week for 8 weeks.
  Other Names: Music Therapy
  Arms: Study (Music) Group

SUMMARY:
The main purpose of this study is to investigate the effect of music therapy on the upper extremity functions and quality of life of individuals with Cerebral Palsy (CP). The secondary aim is to investigate the effect of music therapy on the sensory functions of the upper extremity in individuals with CP. Adolescent individuals with hemiparetic CP will participate in this study, and the participants will experience music therapy, which is a scientific intervention approach. If music therapy has a positive effect on upper extremity functions, they will be more active in daily life and their quality of life will increase. In the light of these data to be presented, a contribution will be made to the evidence level of music therapy in the literature and to the content of SP upper extremity rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 6-21
* With upper extremity dysfunction
* MACS score between 2-4,
* According to MAS, spasticity severity ranges from (1+) to (3),
* Individuals diagnosed with hemiparetic Cerebral Palsy who are at a cognitive level that can follow simple instructions during applications and evaluations will be included.

Exclusion Criteria:

* Having another neurological disorder
* Having undergone upper extremity orthopedic surgery or Botulinum Toxin A (BTX-A) application in the last 6 months,
* Individuals currently receiving another rehabilitation program in addition to classical physiotherapy for upper extremity rehabilitation will be excluded from the study.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-17 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Children's Hand-Use Experience Questionnaire (CHEQ) | Change from baseline at 8 weeks
  Children's Hand-Use Experience Questionnaire (CHEQ) is a scale that evaluates unilateral hand disorders in children due to various reasons (such as hemiparetic CP, brachial plexus or upper extremity developmental deficiency for any reason). CHEQ consists of 27 sub-items and evaluates quality aspects of movement in three different subscales, including the grasping efficiency of hand functions, the time required to perform the activity, and the feeling of discomfort caused by the affected hand during the performance of the activity.
Abilhand-Kids | Change from baseline at 8 weeks
  Abilhand-Kids scale evaluates hand functions in children with CP. It measures the use of the upper extremity during children's daily activities in 21 items. There are 3 points in the scoring: 0: cannot be done, 1: difficult, 2: easy.
Selective Control of the Upper Extremity Scale (SCUES) | Change from baseline at 8 weeks
  Selective Control of the Upper Extremity Scale (SCUES) is a measurement tool specifically designed for this area, developed to evaluate selective motor control of the upper extremity. It is a useful evaluation measure that is video-based and implemented in less than 15 minutes. The degree of selective motor control is determined for each joint as "normal selective motor control: 3 points, mildly reduced selective motor control: 2 points, moderately reduced selective motor control: 1 point, no selective motor control: 0 points".
Pediatric Quality of Life Inventory (PedsQL) 3.0 Cerebral Palsy Module | Change from baseline at 8 weeks
  Pediatric Quality of Life Inventory (PedsQL) 3.0 Cerebral Palsy (CP) Module was developed to evaluate CP-specific quality of life areas of children with CP between the ages of 2-18. The scale questions the degree of problems experienced by individuals in the last month. The 35-item module consists of seven subscales: daily activities (9 items), school activities (4 items), movement and balance (5 items), pain and suffering (4 items), fatigue (4 items), eating activities (5 items), speech and communication (4 items). Subscale scores are calculated by dividing the total score of the answered items by the number of answered items. A higher mean score on a subscale of a field indicates that there are fewer problems in that field and the quality of life is higher.

SECONDARY OUTCOMES:
Semmes Weinstein Monofilament Test (SWMT) | Change from baseline at 8 weeks
  Semmes Weinstein Monofilament Test (SWMT) is a tactile test battery recommended to evaluate tactile sensation in individuals with CP. The SWMT battery has five different thicknesses of monofilament ranging from 2.83 to 6.65. The evaluation starts with the thinnest (2.83) filament and continues until the monofilament that the individual begins to feel.
Two-Point Discrimination | Change from baseline at 8 weeks
  Two-Point Discrimination is used to evaluate tactile perception in individuals with CP. It evaluates the ability to perceive and distinguish tactile stimuli applied from two different points at the same time. The evaluation starts from the widest gap (15 mm) and progresses to the narrowest gap (0 mm). The lowest distance range that the individual feels is recorded.
Modified Ashworth Scale (MAS) | Change from baseline at 8 weeks
  Modified Ashworth Scale (MAS) is a test that evaluates the increase in muscle tone resulting from increased resistance during passive movement of the extremity. It is a 6-level spasticity measurement method scored in the range of 0-4. The higher the score, the greater the spasticity.

OTHER OUTCOMES:
The Gross Motor Function Classification System (GMFCS) | Before the start of treatment
  The Gross Motor Function Classification System (GMFCS) determines the level most appropriate to an individual's limitations and skills in gross motor functions. This classification measures the individual's self-initiated movements based on displacement, sitting and mobility, regardless of the individual's motor disorder type. As a result of the findings, individuals are divided into 5 levels according to their motor function levels. Individuals at Level 1 have minimal motor limitations.
The Manual Ability Classification System (MACS) | Before the start of treatment
  The Manual Ability Classification System (MACS) classifies how individuals with CP use their hands when holding objects in their daily activities in five levels. The individual at level 1 can hold and use objects easily and successfully, while the individual at level 5 cannot hold and use objects and has extremely limited skills to perform even simple activities. When determining levels, the ability of individuals to hold objects by themselves and the need for assistance in performing manual activities in daily life are taken into account.

CONTACTS AND LOCATIONS:
Overall Officials: Sena ÇARIKCI, MSc, Principal Investigator — Ankara Yıldırım Beyazıt University Health Sciences Institute; Nezehat Özgül ÜNLÜER, PhD, Study Chair — Saglik Bilimleri Universitesi; Şükrü TORUN, MD, Study Chair — Anadolu University Health Sciences Institute
Locations (1):
- Sena ÇARIKCI, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No